CLINICAL TRIAL: NCT03793400
Title: Long-term Outcome of Punctate Inner Choroidopathy or Multifocal Choroiditis With Active Choroidal Neovascularization Managed With Anti-vascular Endothelial Growth Factor
Status: Completed | Type: Observational
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, San Ni Chen, Department of Ophthalmology, Changhua Christian Hospital
Other Study IDs: 180916
Record Dates: First submitted 2019-01-01; First posted 2019-01-04 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Choroidal Neovascularization; Punctate Inner Choroidopathy
Keywords: punctate inner choroidopathy; multifocal choroidits; choroidal neovascularization; anti-VEGF; long-term outcome
MeSH Terms: conditions — Choroidal Neovascularization; White Dot Syndromes | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bevacizumab Injection — Anti-vascular endothelial growth factor (VEGF)

SUMMARY:
To evaluate the long-term outcome of active choroidal neovascularization (CNV) in punctate inner choroidopathy (PIC) or multifocal choroiditis (MFC) after anti-vascular endothelial factor treatment.

DETAILED DESCRIPTION:
To evaluate the long-term outcome of active choroidal neovascularization (CNV) in punctate inner choroidopathy (PIC) or multifocal choroiditis (MFC) after anti-vascular endothelial factor treatment.

The age, sex, best corrected visual acuity (BCVA) in Snellen chart, and refractive status for each patient were recorded. All patients had thorough clinical examinations, including slit lamp biomicroscopy, indirect ophthalmoloscopy, and spectral domain optical coherence tomography during each visit. Fundus photography, fluorescein angiography, and indocyanine angiography were performed on all patients. OCT angiography was performed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were punctate inner choroidopathy or multifocal choroiditis with active choroidal neovascularization.
2. Follow up over 4 years.

Exclusion Criteria:

1. Patients were not punctate inner choroidopathy or multifocal choroiditis with active choroidal neovascularization
2. Patients were punctate inner choroidopathy or multifocal choroiditis with active choroidal neovascularization but loss follow over 1 year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators included punctate inner choroidopathy or multifocal choroiditis with active choroidal neovascularization patients with follow up over 4 years.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Wilcoxon Signed-Rank test | Baseline,48 month.
  A statistical comparison of average of two dependent samples

SECONDARY OUTCOMES:
visual acuity | Baseline,48 month.
  visual acuity in logMAR

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided